CLINICAL TRIAL: NCT04534478
Title: Randomized, Open, Parallel, Single-center, Non-inferiority Clinical Trial, With an Active Control Group, Comparing Two Oral Prednisone Regimens With the Aim of Optimizing the Therapeutic Strategy in Patients With Organizing Pneumonia Post-COVID-19 Infection
Brief Title: Oral Prednisone Regimens to Optimize the Therapeutic Strategy in Patients With Organizing Pneumonia Post-COVID-19
Acronym: NORCOVID
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003651-15
Record Dates: First submitted 2020-08-31; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Parallel clinical trial with therapeutic intervention, randomized, open and controlled, of non-inferiority
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Prednisone 0.75mg / Kg / d 4 weeks; 0.5mg / Kg / d 4 weeks; 20mg / d 4 weeks; 10mg / d 6 weeks; 5mg / d 6 weeks (6m)
  Interventions: Drug: Prednisone
- Experimental group (Active Comparator): Prednisone 0.5mg / Kg / d 3 weeks, 20mg / day 3 weeks; 15mg / day 2 weeks; 10mg / day 2 weeks, 5mg / day 2 weeks and discontinue.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Patients will be randomized 1: 1 between the two arms of the study

SUMMARY:
Background: Based on data from the 2003 SARS-COVID pandemic, other serious lung infections, and patients with respiratory distress, it is estimated that 10-30% of patients with severe SARS-COVID-2 pneumonia may present as a sequel an organized pneumonia. The treatment of this complication is not well defined. The use of oral corticosteroids is mandatory to avoid a possible evolution to pulmonary fibrosis, however, the doses to be administered and the duration of treatment are unknown as there is no study specifically aimed at solving this doubt. Many authors advocate high-dose treatment regimens for a minimum of six months, as proposed for cryptogenic organized pneumonia. However, there is a question whether in non-idiopathic cases of organized pneumonia, less intense treatment could resolve the disease. Hypothesis: The use of a less intensive prednisone regimen may be sufficient for therapeutic control in patients with post-COVID-19 organizing pneumonia, in relation to the established standard regimen Simplicity of the procedures: The objective of the NORCOVID study is to identify the optimal treatment regimen with corticosteroids in post-COVID19 patients diagnosed with NO. Specifically, the primary objective of this multicenter randomized trial is to evaluate whether treatment with a less intensive regimen of corticosteroids produces a non-inferior therapeutic effect than the established control regimen. Secondary objectives are to evaluate the effect of treatment on secondary efficacy variables and on safety. DLCO, respiratory function tests, 6MWT test, need for rescue, radiological tests, complications, mortality and the WHO ordinal scale will be evaluated.

DETAILED DESCRIPTION:
Hypothesis The use of a less intensive prednisone regimen may be sufficient for therapeutic control in patients with post-COVID-19 organizing pneumonia, in relation to the established standard regimen.

Objectives The objective of the NORCOVID study is to identify the optimal treatment regimen with corticosteroids in post-COVID19 patients diagnosed with NO. Specifically, the primary objective of this multicenter randomized trial is to evaluate whether treatment with a less intensive regimen of corticosteroids produces a non-inferior therapeutic effect than the established control regimen. Secondary objectives are to evaluate the effect of treatment on secondary efficacy variables and on safety. DLCO, respiratory function tests, 6MWT test, need for rescue, radiological tests, complications, mortality and the WHO ordinal scale will be evaluated.

Study population: inclusion and exclusion criteria

* Inclusion criteria 1) Patients over 18 years of age 2) Diagnosis of COVID-19 pneumonia that would have required hospital admission 3) Diagnosis of post-COVID-19 organized pneumonia 4) Without any contraindication to the study drug 5) That, properly informed, voluntarily agree to participate in the study after knowing its objectives and risks and give their consent.
* Exclusion criteria Patients will not be randomized if: 1) They do not authorize their participation 2) Patients with contraindications to receiving corticosteroid treatment 3) Impossibility of understanding the requirements of the study, in the opinion of the investigator. 4) Expected survival less than the duration of the study in the opinion of the investigator. 5) Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis, urinary tract infection, and / or cellulitis. 6) Patient who is subject to receiving a lung transplant during the study period. 7) Impossibility of conducting lung function studies. 8) Poorly controlled diabetes mellitus (glycosylated Hb> 10%). 9) Pregnancy or breastfeeding 10) Have any contraindication to the study drug 11) Are participating in another intervention study.

Products evaluated and administration regimens.

The product evaluated will be Prednisone orally in two administration schedules:

1. Control Group: Prednisone 0.75mg / Kg / d 4week; 0.5mg / Kg / d 4 weeks; 20mg / d 4 weeks; 10mg / d 6 weeks; 5mg / d 6 weeks (6m).
2. Experimental Group: Prednisone 0.5mg / Kg / d 3 weeks, 20mg / day 3 weeks; 15mg / day 2 weeks; 10mg / day 2 weeks, 5mg / day 2 weeks and discontinue.

Main variable - The main variable will be the change in pulmonary diffusion, in terms of predicted DLCO (%), between the baseline value and that obtained at 6 months, comparing the two treatment groups adjusting for the baseline value using a model of Repeated measures with random effects (mixed model for repeated measurements: MMRM).

Secondary variables

* DLCO in original units (DLCO10s mLmin - 1mmHg - 1)
* Percentage of patients with values <80% predicted
* Respiratory function tests
* 6-Minute-Walk Test (6MWT) test
* Need for rescue
* Computed Axial Tomography Test
* Complications related to the evolution of the disease (serious and non-serious)
* Complications related to corticosteroid treatment (serious and non-serious)
* Complication of any kind (serious and non-serious)
* Mortality from any cause
* Ordinal variable of clinical improvement recommended by the WHO R&D Blueprint expert group15 for the acute phase. The worst score obtained during the study will be evaluated at each visit and as a summary measure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Diagnosis of COVID-19 pneumonia that would have required hospital admission
* Post COVID-19 Organized Pneumonia Diagnosis
* Without any contraindication to the study drug
* That, adequately informed, voluntarily agree to participate in the study after knowing its objectives and risks and grant their written consent.

Exclusion Criteria:

* They do not authorize their participation
* Patients with contraindications to receiving treatment with corticosteroids
* Impossibility of understanding the requirements of the study, in the opinion of the researcher.
* Expected survival less than the duration of the study in the opinion of the investigator.
* Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis, urinary tract infection and / or cellulitis.
* Patient who receives a lung transplant during the study period.
* Impossibility of carrying out lung function studies. - Poorly controlled diabetes mellitus (glycosylated Hb> 10%).
* Pregnancy or breastfeeding
* They are participating in another intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-07 (Estimated); Primary Completion 2021-05-02 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary diffusion. | Six Months
  The main variable will be the change in pulmonary diffusion, in terms of predicted DLCO (%), between the baseline value and that obtained at 6 months, comparing the two treatment groups, adjusting for the baseline value using a repeated measures model with random effects (mixed model for repeated measurements.

IPD SHARING:
Plan to Share IPD: No